CLINICAL TRIAL: NCT03828149
Title: Evaluation of Safety and Pharmacodynamics of OP0201 Compared to Placebo
Brief Title: Evaluation of Safety and Pharmacodynamics of OP0201 Compared to Placebo in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novus Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: OP0201-C-001
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-10

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug: OP0201 (Active Comparator): 20 mg dose one time, followed by a washout and then a 0 mg dose one time, cross over design
  Interventions: Combination Product: Drug:OP0201
- Drug: Placebo (Placebo Comparator): 0 mg dose one time, followed by a washout and then a 20 mg dose one time, cross over design
  Interventions: Combination Product: Drug: Placebo

INTERVENTIONS:
Combination Product: Drug:OP0201 — Drug: OP0201
  Arms: Drug: OP0201
Combination Product: Drug: Placebo — Drug: Placebo
  Arms: Drug: Placebo

SUMMARY:
Evaluation of Safety and Pharmacodynamics of OP0201 Compared to Placebo in Healthy Adults

DETAILED DESCRIPTION:
Evaluation of Safety and Pharmacodynamics of OP0201 Compared to Placebo in Healthy Adults

ELIGIBILITY:
Inclusion Criteria includes but is not limited to:

1. Body Mass Index (BMI) 18 to 30 and a minimum body weight of 50 kg at screening.
2. No history or presence of significant medical condition or a clinically significant abnormal finding, as determined by the investigator.
3. Negative urine pregnancy test at screening and baseline for females of childbearing potential
4. Agree to refrain from water immersion of the ears from the time of signed informed consent to the end of trial
5. Physiologic tympanogram type A (normal) or type C at screening visit

Exclusion Criteria includes but is not limited to:

1. Known substance abuse (e.g., alcohol, licit or illicit drugs) within 96 weeks prior to screening visit
2. Positive urine drug screen at screening visit
3. Upper respiratory tract infection currently or within 6 weeks prior to screening visit
4. Allergy or sinus conditions (e.g., sinusitis, non-specific nasal inflammation) currently or within 6 weeks prior to screening visit
5. Claustrophobia that is sufficient to prevent them tolerating assessments while in a hypobaric/hyperbaric atmospheric pressure chamber
6. Smoker (e.g ., cigarettes, vapor) within the last 48 weeks prior to screening visit
7. Clinically significant findings on ear nose and throat exam
8. Gastroesophageal reflux disease currently or within 6 weeks prior to screening visit
9. Current diagnosis of sleep apnea
10. Evidence of craniofacial anomalies (eg, cleft palate, Down's Syndrome) that may interfere with ET function
11. Disorders with decreased mucociliary clearance or higher viscosity of the mucous (eg, cystic fibrosis, primary ciliary dyskinesia, Kartagener's syndrome)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cologne University Hospital, Cologne, Germany

REFERENCES:
- See also: Related Info — http://novustherapeutics.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: OP0201 First, Then Placebo: Participants first received 20mg one time dose of OP0201, followed by a washout and then a single dose of Placebo, cross over design
  Drug:OP0201: Drug: OP0201
- Drug: Placebo First, Then OP0201: Participants first received 0 mg one time dose of Placebo, followed by a washout and then a single dose of OP0201, cross over design
  Drug: Placebo: Drug: Placebo
Period: First Intervention (Single Dose)
Arm/Group | Drug: OP0201 First, Then Placebo | Drug: Placebo First, Then OP0201
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0
Period: Washout (6 Days)
Arm/Group | Drug: OP0201 First, Then Placebo | Drug: Placebo First, Then OP0201
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0
Period: Second Intervention (Single Dose)
Arm/Group | Drug: OP0201 First, Then Placebo | Drug: Placebo First, Then OP0201
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Drug: OP0201 First, Then Placebo: Participants first received 20mg one time dose, followed by a washout and then a single dose of the opposite intervention, cross over design
  Drug:OP0201: Drug: OP0201
- Drug: Placebo First, Then OP0201: Participants first received 0 mg one time dose, followed by a washout and then a single dose of the opposite intervention, cross over design
  Drug: Placebo: Drug: Placebo
- Total: Total of all reporting groups
Arm/Group | Drug: OP0201 First, Then Placebo | Drug: Placebo First, Then OP0201 | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (5.7) | 24.5 (3.9) | 25.8 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety (Evaluation of Adverse Events)
Description: All randomized participants who received at least one spray of study treatment in either nare were included in the safety analysis.
Time Frame: Days 1-9
Measure: Count of Participants; unit: Participants
Groups:
- Drug: OP0201: Participants received 20mg OP0201 one time dose at Day 1 or Day 8.
  Drug:OP0201: Drug: OP0201
- Drug: Placebo: Participants received 0 mg one time dose at Day 1 or Day 8.
  Drug: Placebo: Drug: Placebo
Arm/Group | Drug: OP0201 | Drug: Placebo
Number analyzed (Participants) | 17 | 17
Participants | 17 | 17

ADVERSE EVENTS:
Time Frame: 9 days
Description: The safety population included all randomized participants who received at least one spray of study treatment in either nare.
Groups:
- OP0201: Participants received OP0201 20mg one time dose at either Day 1 or Day 8.
  Drug:OP0201: Drug: OP0201
- Placebo: Participants received Placebo 0 mg one time dose at either Day 1 or Day 8.
  Drug: Placebo: Drug: Placebo
Arm/Group | OP0201 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 12/17 | 14/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OP0201 (N=17) | Placebo (N=17)
Ear Pain (Ear and labyrinth disorders) | 8 | 10
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 6 | 5
Tympanic membrane disorder (Ear and labyrinth disorders) | 4 | 3
Ear discomfort (Ear and labyrinth disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 4
Dizziness (Nervous system disorders) | 1 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT03828149/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT03828149/SAP_001.pdf